CLINICAL TRIAL: NCT02884336
Title: Lactobacillus Plantarum: Thumb Osteoarthritis Following Orange Peeling
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Lactobacillus plantarum
Record Dates: First submitted 2016-07-20; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Lactobacillus Plantarum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
Case Description osteoarthritis + amputation of the distal phalanx of the right thumb caused by Lactobacillus plantarum after an orange peel. The natural habitat of the bacteria being the orange zest and the bacteria is considered harmless.

DETAILED DESCRIPTION:
Case Description osteoarthritis + amputation of the distal phalanx of the right thumb caused by Lactobacillus plantarum after an orange peel. The natural habitat of the bacteria being the orange zest and the bacteria is considered harmless.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an osteoarthritis,
* Amputation of the distal phalanx of the right thumb

Exclusion Criteria:

* Not exclusion criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A patient who had osteoarthritis + amputation of the distal phalanx of the right thumb caused by Lactobacillus plantarum after an orange peel.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Identification of Lactobacillus plantarum | Day 1
  This study was conducted like a case report to describe osteoarthritis + amputation of the distal phalanx of the right thumb caused by Lactobacillus plantarum after an orange peel. The natural habitat of the bacteria being the orange zest and the bacteria is considered harmless

CONTACTS AND LOCATIONS:
Overall Officials: Mizrahi Assaf, Assaf, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France